CLINICAL TRIAL: NCT01682967
Title: Alteration in Hearing Following Accidental Dural Puncture. A Study in Parturients
Acronym: AHEAD
Status: Completed | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Other Study IDs: AHEAD-11
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Parturients in Labour
Keywords: Parturients; Analgesia, epidural; Headache, post-dural puncture
MeSH Terms: conditions — Agnosia; Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Experimental group: Patients suffering from PDPH would form this group
- Control group - Epidural: Patients who received an epidural during labour but did not have symptoms of PDPH would form this reference group
- Control Group without Epidural analgesia: Patients in labour who did not receive an EDA would form this cohort of controls

SUMMARY:
Headache following accidental dural punction as during epidural analgesia can be severe and sometimes very disabling. The incidence of PDPH is 10-40%, most starting within 48 h of dural puncture. Although spontaneous resolution of headaches is common in most patients within 7 days, in 20% can they be persistent and in some very disabling. The exact reason for the characteristic headache is unknown, but it is believed to be the result of leakage of cerebro-spinal fluid (CSF) from the dural puncture. The greater the leakage of CSF, the more severe and persistent the headache. This is why larger needles (lower gauge) are known to have a higher incidence of PDPH. However, the type of needle also seems to play an important role in the likelihood of PDPH.

Headache following accidental PDPH is very typical as it increases significantly when sitting or standing and often disappears completely on lying down. It is typically located in the back of the head, accentuated by light and often decreases with intake of large quantity of fluids. In many cases, it is self-limiting and most often decreases with time and bed rest.

Diagnosis of PDPH is clinical and sometimes difficult. It is well known that liquor leakage, as following spinal anaesthesia, results in partial loss of unilateral or bilateral hearing that can be detected by oto-acoustic hearing loss. We plan to use this knowledge and test the hypothesis that measurement of hearing loss may be a diagnostic method for confirmation of clinical symptoms and signs of accidental PDPH.

DETAILED DESCRIPTION:
Parturients who have received epidural analgesia during labour would be included in this study and these would comprise of:

1. patients without clinical symptoms of postdural puncture headache
2. patients with clinical symptoms of postdural puncture headache

In addition, a control group of parturients who have not received an epidural analgesia would constitute the control group.

All patients would have audiometry (oto-acoustic emission - OAE, and auditory steady state response - ASSR) done following diagnosis of PDPH. Subsequently, the patients would be observed for 24 h to assess whether the headache resolves spontaneously. A new audiometry would be done at this stage. Those patients with substantial evidence of PDPH at this stage would receive an epidural blood patch (EBP) and a new audiometric assessment would be made after 4 h and 24 h to assess whether any audiometric deficit has resolved or not. All patients would have a similar measurement of hearing after 3 months when it is believed that most patients have returned to normal hearing. In addition to audiometric analysis, patients would be asked to fill out a detailed PDPH questionnaire at the same time periods.

All measurements would be compared with patients who have received an EDA but without PDPH and those who have not received an EDA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy parturients No known hearing problems Understand Swedish language Informed consent

Exclusion Criteria:

* Taking steroid medication Having pre-eclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Experimental group: Parturients in labour with epidural and having PDPH Control group - EDA: Parturients in labour with epidural and NOT having PDPH Control group - No EDA: Parturients in labour without epidural and NOT having PDPH
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post-dural puncture headache | 4 h after epidural blood patch
  VAS pain (headache) 4 h after application of EBP

SECONDARY OUTCOMES:
Audiometric data | 4 h following EBP
  OAE and ASSR would be measured 4 h after application of EBP
PDPH questionnaire | 4 h after application of EBP
  The PDPH questionnaire would be used to analyse pain and its characteristics 4 h after application of EBP
Recurrence of Headache | 24 h after application of EBP
  The incidence of recurrence of PDPH after initial improvement on application of EBP would be recorded after 24 h

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - University Hospital, Örebro
  - Karolinskasjukhuset, Solna